CLINICAL TRIAL: NCT06586944
Title: After the Research Groups Were Formed, a Six-session Interview Program Was Created for the Participants Included in the Experimental Group. During These Sessions, Nursing and Psychiatric Nursing Interventions (psychoeducation, Relaxation, Awareness, Effective Coping, Cognitive Restructuring) Based on RAM Were Conducted to Address the Negative Situations Caused by Anxiety and Anxiety Experienced by Individuals. Subjective Goals Were Determined for the Adaptive or Maladaptive Behavior, Attitude, and Thought Patterns Caused by the Anxiety-causing Stimuli.
Brief Title: Effect of Nursing Interventions Using Roy Adaptation Model with Virtual Reality on Social Anxiety in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aytuğ Türk (Other)
Collaborators: Aliye Üster Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Aytuğ Türk, Research Asistant, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ATurk
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Social Anxiety Disorder
Keywords: social anxiety; young people; Roy Adaptation Model; virtual reality; psychiatric nursing
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: After the research groups were formed, a six-session interview program was created for the participants included in the experimental group. During these sessions, nursing and psychiatric nursing interventions (psychoeducation, relaxation, awareness, effective coping, cognitive restructuring) based on RAM were conducted to address the negative situations caused by anxiety and anxiety experienced by individuals.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group (Experimental): After the research groups were formed, a six-session interview programme was created for the participants included in the experimental group . In the sessions, nursing and psychiatric nursing interventions (psychoeducation, relaxation, awareness, effective coping, cognitive restructuring) based on the Roy Adaptation Model were carried out for the negative situations caused by anxiety and anxiety experienced by individuals. Virtual reality-based intervention was effectively used as an important intervention tool in the implementation of the interventions and in the evaluation of the implemented interventions in four sessions of a total of six sessions. During the application, the participants were asked to evaluate their anxiety in the range of 0-10 as subjective feedback via the 'Amelia VR Platform', and ratings were requested every three minutes during the 15-minute experience of the virtual reality platform, especially at moments when their anxiety increased subjectively.
  Interventions: Behavioral: Nursing Practices Based On Roy Adaptation Model Integrated With Virtual Reality
- Control Group-2 (No Intervention): No intervention was made to the participants in the II. Control group except for the completion of the pre-test, post-test and follow-up test.
- Control Group (Active Comparator): For the participants in the control group, a six-session interview programme was created in a way that virtual reality application was not used. In the sessions, nursing and psychiatric nursing interventions (psychoeducation, relaxation, awareness, effective coping, cognitive restructuring) based on the Roy Adaptation Model were carried out for the negative situations caused by anxiety and anxiety experienced by individuals. Subjective goals were determined for the adaptive or maladaptive behaviour, attitude and thought patterns caused by anxiety-inducing stimulus(s) and appropriate interventions from the Nursing Interventions Classification System (NIC) were carried out for these goals.
  Interventions: Behavioral: Roy Adaptation Model

INTERVENTIONS:
Behavioral: Nursing Practices Based On Roy Adaptation Model Integrated With Virtual Reality — After the research groups were formed, a six-session interview programme was created for the participants included in the experimental group (Table...). In the sessions, nursing and psychiatric nursing interventions (psychoeducation, relaxation, awareness, effective coping, cognitive restructuring) based on the Roy Adaptation Model were carried out for the negative situations caused by anxiety and anxiety experienced by individuals. Subjective goals were determined for adaptive or maladaptive behaviour, attitude and thought patterns caused by anxiety-causing stimulus(s) and appropriate nursing interventions from the Nursing Interventions Classification System (NIC) were applied for these goals.Virtual reality-based intervention was effectively used as an important intervention tool in the implementation of the interventions and in the evaluation of the implemented interventions in four sessions of a total of six sessions.
  Arms: Experimental group
Behavioral: Roy Adaptation Model — After the research groups were formed, a six-session interview programme was created for the participants included in the experimental group. In the sessions, nursing and psychiatric nursing interventions (psychoeducation, relaxation, awareness, effective coping, cognitive restructuring) based on the Roy Adaptation Model were carried out for the negative situations caused by anxiety and anxiety experienced by individuals. Subjective goals were determined for adaptive or maladaptive behaviour, attitude and thought patterns caused by anxiety-causing stimulus(s) and appropriate nursing interventions from the Nursing Interventions Classification System (NIC) were applied for these goals
  Arms: Control Group

SUMMARY:
The study was conducted to determine the effect of nursing practices based on the RAM integrated with VR on the social anxiety level of young people.The main questions it aims to answer are:

H1: "Nursing practices based on the Roy Adaptation Model integrated with virtual reality are effective in reducing the level of social anxiety in young people." H2: "Nursing practices based on the Roy Adaptation Model integrated with virtual reality are effective on the level of life satisfaction, independent of anxiety level and as a predictor of social anxiety"

This single-blinded randomized controlled study utilized a pretest-posttest control group and single-blinded randomized control group, preintervention pretest, postintervention posttest, and follow-up test design. The study population consisted of students from a foreign language preparatory class at a university. In this context, the Anxiety Subdimension of the LSCQ was calculated for 785 preparatory class students aged 18-26. A total of 242 students scoring 30 and above on the Anxiety Subdimension of the LSCQ were reached. The research was completed with a sample of 72 students who met the inclusion criteria within this target group. Individuals who do not participate in two or more of the six interviews will be excluded from the study. The study's experimental design was organized according to the CONSORT guidelines

DETAILED DESCRIPTION:
The study used virtual environments and characters based on "The Amelia VR Platform" for mental health researchers developed by Psious software company as a supportive tool in nursing interventions for social anxiety. The virtual environments included scenarios such as presentating in a large conference hall, conducting a business/office meeting with an authority figure and colleagues, presenting to a small group in a seminar hall, and socializing with friends. These environments comprehensively evaluate individuals' issues in public speaking and can also be used within the scope of a separate program to test and improve skills such as verbal communication and academic presentation. The whole process is controlled by a counselor via a computer connected to the platform. The counselor can manipulate the content, duration, and intensity of the process in a controlled manner for the purpose of the application.

ELIGIBILITY:
Inclusion Criteria:

* Liebowitz Social Anxiety Scale (LSAS) anxiety subscale score of 30 and above,
* Having not used a psychiatric drug in the last three months,
* Not having received psychotherapy for social anxiety before,
* Willingness and volunteering to participate in the research.

Exclusion Criteria:

* Active suicide risk,
* Psychotic symptoms,
* Individuals who do not participate in two or more of the six interviews will be excluded from the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Social Anxiety Scale Scores | 3 Months
  Measurement of the change in Social Anxiety Scale Scores Liebowitz Social Anxiety Scale (LSAS) and Satisfaction with Life Scale (SWLS) were reapplied to the experimental and control groups as post-test measurement tools after the intervention and six-week follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The Complete Study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Indefinite Duration
Access Criteria: Since the study is a doctoral thesis, people who want to access the full study can access the study in the database of the Council of Higher Education of Turkey (YÖK).
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp